CLINICAL TRIAL: NCT02127515
Title: Non Invasive Prenatal Testing of Down Syndrome From Maternal Blood Sample
Brief Title: Non Invasive Prenatal Testing of Down Syndrome
Acronym: SAFE 21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P130601; 2013-A00998-37 (Other: ANSM)
Record Dates: First submitted 2014-04-02; First posted 2014-04-30 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Down Syndrome
Keywords: Down, trisomy 21; NIPT; Amniocentesis; miscarriage; invasive; prenatal; screening.
MeSH Terms: conditions — Down Syndrome; Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non Invasive Prenatal Testing (Experimental): Blood sample
  Interventions: Procedure: Non Invasive Prenatal Testing
- Invasive Prenatal Testing (Active Comparator): CVS or amniocentesis
  Interventions: Procedure: Invasive Prenatal Testing

INTERVENTIONS:
Procedure: Non Invasive Prenatal Testing
  Arms: Non Invasive Prenatal Testing
Procedure: Invasive Prenatal Testing
  Arms: Invasive Prenatal Testing

SUMMARY:
This is a randomized controlled trial in women at risk following combined prenatal screening for Down Syndrome. Women will be asked about their preferences between NIPT and routine prenatal diagnosis based on a dedicated questionnaire. Women will then be randomized between NIPT and standard invasive prenatal diagnosis.

DETAILED DESCRIPTION:
This is a randomized controlled trial in women at risk following combined prenatal screening for Down Syndrome. Women will be asked about their preferences between NIPT and routine prenatal diagnosis based on a dedicated questionnaire. Women will then be randomized between NIPT and standard invasive prenatal diagnosis.

The general objectives are :

* Promote the rapid and large implementation of Non Invasive Prenatal Testing (NIPT) for Down syndrome.
* Improve the management of women at risk after combined first trimester screening and reduce the number of invasive procedures and induced miscarriages .
* Evaluate NIPT medically (in reducing the rate of invasive sampling and related complications, diagnostic performance and feasibility and acceptability in routine practice) and based on cost-analysis in comparison with standard invasive prenatal diagnosis currently proposed .
* Clarify the conditions of implementation and dissemination of NIPT in the overall organization of prenatal screening for trisomy 21 (and provide data to later adjust or not the combination of tests and thresholds).

Promote the organization as networks of professionals involved in prenatal screening for trisomy 21 in order to allow the emergence of a national system of collection of outcomes to improve the quality of practices

The main judgement criteria are:

* Main:

  - Percentage of fetal loss in each group
* Secondary:

  * Percentage of invasive tests in each group (amniocentesis or chorionic villus sampling )
  * Diagnostic performance of NIPT , in particular false positive and negative
  * Percentage of results within 3 weeks and average time interval for results of NIPT
  * Percentage of inconclusive results of DPANI
  * Percentage of other anomalies discovered at invasive sampling
  * Percentage of invasive samples taken despite normal NIPT (either because of later ultrasound anomaly or for maternal reinsurance)
  * Association between maternal characteristics ( weight, height, parity , previous history , serum markers ... ) and the results of NIPT
  * Cost analysis of NIPT in routine clinical practice

The study will include 2450 high risk women in order to be powered enough to detect a 1% reduction of miscarriages in the group undergoing NIPT instead of routine invasive prenatal diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women over 18
* at risk for Down syndrome> 1/250 based on combined screening using ultrasound together with maternal serum markers and prior to fetal karyotyping
* singleton pregnancy
* pregnancy between 11SA et 18SA
* willing a fetal karyotype

Exclusion Criteria:

* risk for Down syndrome< 1/250 or >1/5
* NT> 3 mm, PAPP-A or beta HCG <0.3 MoM or >5 MoM
* multiple pregnancy , vanishing twin
* morphological abnormalities at US
* Kown chromosomal anomaly in parents
* Patients not willing a fetal karyotype

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2111 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2016-11-07 (Actual)

PRIMARY OUTCOMES:
Number or miscarriages | at birth

SECONDARY OUTCOMES:
Number or invasive tests | at birth
false positive and negative rates of NIPT | At birth
Dedicated questionnaire for patients | day 5
Cost of invasive tests and NIPT in euros | at birth
  measure in euros

CONTACTS AND LOCATIONS:
Overall Officials: Laurent J Salomon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Michel VEKEMANS, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker- Enfants Malades, Paris, France

REFERENCES:
- [Background] Le Bras A, Salomon LJ, Bussieres L, Malan V, Elie C, Mahallati H, Ville Y, Vekemans M, Durand-Zaleski I. Cost-effectiveness of five prenatal screening strategies for trisomies and other unbalanced chromosomal abnormalities: model-based analysis. Ultrasound Obstet Gynecol. 2019 Nov;54(5):596-603. doi: 10.1002/uog.20301. PMID 31006923
- [Background] Seror V, L'Haridon O, Bussieres L, Malan V, Fries N, Vekemans M, Salomon LJ, Ville Y; SAFE 21 Study Group. Women's Attitudes Toward Invasive and Noninvasive Testing When Facing a High Risk of Fetal Down Syndrome. JAMA Netw Open. 2019 Mar 1;2(3):e191062. doi: 10.1001/jamanetworkopen.2019.1062. PMID 30924894
- [Background] Malan V, Bussieres L, Winer N, Jais JP, Baptiste A, Le Lorc'h M, Elie C, O'Gorman N, Fries N, Houfflin-Debarge V, Sentilhes L, Vekemans M, Ville Y, Salomon LJ; SAFE 21 Study Group. Effect of Cell-Free DNA Screening vs Direct Invasive Diagnosis on Miscarriage Rates in Women With Pregnancies at High Risk of Trisomy 21: A Randomized Clinical Trial. JAMA. 2018 Aug 14;320(6):557-565. doi: 10.1001/jama.2018.9396. PMID 30120476